CLINICAL TRIAL: NCT03320304
Title: A Global PRospective, Multi-cEnter, ObServational Post-markeT Study tO Assess shoRt, Mid and Long-term Effectiveness and Efficiency of VNS Therapy® as Adjunctive Therapy in reaL-world patIents With diFficult to Treat dEpression.
Brief Title: A Study to Assess Effectiveness and Efficiency of VNS Therapy in Patients With Difficult to Treat Depression.
Acronym: RESTORE-LIFE
Status: Recruiting | Type: Observational
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Other Study IDs: LNN800
Record Dates: First submitted 2017-10-05; First posted 2017-10-25 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Treatment Resistant Depression
Keywords: Difficult to Treat Depression; TRD; VNS Therapy; Vagus Nerve Stimulation; VNS
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Vagal Nerve Simulation (VNS) Therapy: The aim of this study is to include patients with difficult to treat depression from a global "real world" (standard of care) population who are referred for treatment with VNS Therapy.
  Interventions: Device: Vagal Nerve Simulation (VNS) Therapy

INTERVENTIONS:
Device: Vagal Nerve Simulation (VNS) Therapy — A VNS Therapy System used for vagus nerve stimulation and consisting of an implantable VNS Therapy generator, lead, and external programming system.

SUMMARY:
The primary objective of this study is to assess short, mid and long-term clinical outcomes in patients with difficult to treat depression (such as patients with treatment resistant depression) treated with Vagus Nerve Stimulation (VNS) Therapy as adjunctive therapy.

DETAILED DESCRIPTION:
The population under study comprises a real-world patient population with difficult to treat depression: patients diagnosed with unipolar or bipolar disorder with chronic or recurrent depression who fail to achieve an adequate response to standard psychiatric management.

The diagnosis of depression and comorbid disorders will be determined based on the Mini International Neuropsychiatric Interview (MINI).

A minimum of five hundred (500) patients will be implanted with a VNS Therapy System and up to eighty (80) sites may participate in this study.

Enrollment will take 8 years, based on competitive enrollment. For each subject a baseline visit will occur between 1 and 6 weeks before implant.

Once implanted with the device, subjects will be followed-up for a minimum of 36 months and a maximum of 60 months. The study may stop when the last subject has reached the 36 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age.
* Have a documented primary diagnosis of chronic (>2 years) or recurrent (2 or more prior episodes) major depressive episode that has not adequately responded to an adequate number of antidepressant treatments, as per local medical standards. This diagnosis must be confirmed using the MINI.
* Provide written Ethics Committee (EC) or Institutional Review Board (IRB) approved informed consent and Health Insurance Portability and Accountability Act (HIPAA, US only) authorization (as applicable according to local requirements).
* Currently is receiving at least one antidepressant treatment (i.e., antidepressant drug, maintenance electroconvulsive therapy, or formal psychotherapy including supportive psychotherapy) or mood stabilizing treatment for bipolar patients (such as lithium, anticonvulsants, or atypical antipsychotics).
* Able and willing to comply with the frequency of (outpatient) clinic visits and to reliably complete all the evaluations as specified in the study protocol.Hence based on the nature of their disease, the following patients should not be included: patients with mental retardation, current severe or significant substance/alcohol abuse, diagnosis of one or more schizophrenia-spectrum or other psychotic disorders, diagnosis of borderline or severe personality disorder as determined by clinical judgment which, in the investigator's opinion, would significantly interfere with subject's participation in the study)

Exclusion Criteria:

There are no exclusion criteria; the investigator should refer to the (local applicable) VNS Therapy Physician's Manual.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population under study comprises a real-world patient population with difficult to treat depression: patients diagnosed with unipolar or bipolar disorder with chronic or recurrent depression who fail to achieve an adequate response to standard psychiatric management.
  The diagnosis of depression and comorbid disorders will be determined based on the Mini International Neuropsychiatric Interview (MINI).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-12-14 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this study is response defined as reduction in Montgomery Åsberg Depression Rating Scale (MADRS) total score of at least 50% from baseline to 12 months post implant. | 12 months
  MADRS is a 10-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Each item yields a score of 0 to 6. The overall score ranges from 0 to 60. Higher MADRS score indicates more severe depression.
  A 'Responder' is a subject that achieved ≥ 50% reduction from baseline in MADRS total score at the M12 assessment. A 'Non-Responder' is any patient who did not achieve ≥ 50% reduction from baseline in MADRS score at the M12 assessment.
  No formal hypothesis testing is presented; all the proposed statistical tests are descriptive in nature.
  The Primary endpoint analysis as defined above will be done only on patients that are enrolled while in a major depressive episode (MDE); the cut off point for current MDE at time of implant will be a MADRS score of 20.
  For the patients with a MADRS score below 20 at time of enrollment, only the continuous change in MADRS can be described (as the MADRS can only worsen or stay the same).

SECONDARY OUTCOMES:
Duration of response | through study completion, an average of 4 years
  computed as the difference between the first recorded date post baseline that response is achieved (MADRS reduction from baseline ≥ 50%) and the first date at which MADRS again increased to a level of <40% from baseline.
Change in MADRS | through study completion, an average of 4 years
  Change in MADRS over time
Cumulative response | through study completion, an average of 4 years
  Cumulative percentage of first-time MADRS responders (MADRS reduction from baseline ≥ 50%) at any post-baseline visit.
Cumulative remission | through study completion, an average of 4 years
  Cumulative percentage of subjects in remission (MADRS ≤9) at any post-baseline visit.
Changes in depression score As measured by the Quick Inventory of Depressive Symptomatology Self-Report (QIDS-SR). | through study completion, an average of 4 years
  The Quick Inventory of Depressive Symptomatology (QIDS-SR) is a 16-item, subject-completed questionnaire of the symptoms of mood and depression. The total score ranges from 0 to 27. A higher QIDS-SR score indicates a more severe depression.
Changes in mania score as measured by the Altman Self-Rating Mania Scale (ASRM)*. | through study completion, an average of 4 years
  *Optional assessments: to be done at selected sites only and based on investigator's clinical judgment to decide which subjects complete them.
  The Altman Self-rating Mania Scale (ASRM) is a 5-item self-reported diagnostic scale which can be used to assess the presence and severity manic and hypomanic symptoms, most commonly in patients diagnosed with bipolar disorder. The total score ranges from 0 to 20. A score of 6 or higher indicates a high probability of a manic or hypomanic condition.
Changes in Quality of Life as measured by the EuroQol five dimensions questionnaire (EQ-5D-5L) | through study completion, an average of 4 years
  The EuroQol five dimensions questionnaire (EQ-5D-5L) is a standardized 5-item subject completed questionnaire measuring generic health status and quality of life.
Changes in patient function as measured by the Work Productivity and Activity Impairment Scale (WPAI) | through study completion, an average of 4 years
  The Work Productivity and Activity Impairment Questionnaire (WPAI) is a subject self-reported 6-item questionnaire that measures impairments in work and activities. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Changes in Quality of Life and patient function as measured by the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) | through study completion, an average of 4 years
  The Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) is a standardized 16-item, self-report scale to assess the degree of enjoyment and satisfaction experienced by the subject during the past week.
Changes in suicidality as measured by item #10 of MADRS. | through study completion, an average of 4 years
  Item 10 on the Montgomery-Åsberg Depression Rating Scale (MADRS) scale assesses suicidal thoughts as representing the feeling that life is not worth living, that a natural death would be welcome, suicidal thoughts and preparations for suicide and is rated from 0 to 6. A score of ≥ 4 ('probably better off dead') is of particular interest.
Changes in suicidality as measured by item #12 of QIDS-SR. | through study completion, an average of 4 years
  For Item 12 of the Quick Inventory of Depressive Symptomatology (QIDS-SR), the subject assesses any thoughts of death or suicide over the previous 7 days on a 4- point scale; a score of ≥ 2 ('I think of suicide or death several times a week for several minutes') being of interest.
Changes in adjunctive antidepressant pharmacological treatment | through study completion, an average of 4 years
  All adjunctive concomitant antidepressant and psychotropic medications will be collected
Changes in adjunctive antidepressant non-pharmacological treatment | through study completion, an average of 4 years
  The following adjunctive non-pharmacological treatments will be collected: maintenance electroconvulsive therapy (ECT), Transcranial Magnetic Stimulation (TMS) and psychotherapy
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | through study completion, an average of 4 years
  The following adverse events will be collected: serious adverse events, deaths, VNS Therapy related adverse events and device deficiencies.
Changes in cognition | through study completion, an average of 4 years
  As measured by THINC-it® Tool*.
  *Optional assessments: to be done at selected sites only and based on investigator's clinical judgment to decide which subjects complete them.
Changes in anxiety as measured by the Generalized Anxiety Disorder Assessment (GAD 7)*. | through study completion, an average of 4 years
  *Optional assessments: to be done at selected sites only and based on investigator's clinical judgment to decide which subjects complete them.
  The Generalized Anxiety Disorder 7 (GAD-7) is a 7-item self-reported questionnaire for screening and severity measuring of generalized anxiety disorder (GAD). GAD-7 has seven items and uses a normative system of scoring. Assessment is indicated by the total score, which made up by adding together the scores for the scale all seven items.

CONTACTS AND LOCATIONS:
Overall Officials: Koen Demyttenaere, Prof., Principal Investigator — KU Leuven; Allan Young, Prof., Principal Investigator — King's College
Locations (18):
- AKH Allgemeines Krankenhaus der Stadt Wien, Vienna, Austria
- KU Leuven, Leuven, Belgium
- Germany (12):
  - Sozialstiftung Bamberg - Klinikum am Bruderwald, Bamberg
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Köln, Cologne
  - LVR-Hospital Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsmedizin Göttingen, Göttingen
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena, Jena
  - Universitätsklinik Leipzig, Leipzig
  - University Hospital Münster, Münster
  - Klinikum Wilhelmshaven, Wilhelmshaven
- United Kingdom (4):
  - Glenfield hospital, Leicester
  - King's College London, London
  - Academic Psychiatry Wolfson Research Centre, Newcastle upon Tyne
  - Mendip HTT / St Andrew's Ward, Wells

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kavakbasi E, Kraus C, Reif-Leonhard C, Blackwell JM, Dibue M, Treiber M, Achten S, Baune BT. Titration of vagus nerve stimulation for difficult-to-treat depression and onset of response: Early insights from the RESTORE-LIFE study. J Affect Disord. 2025 Jun 1;378:39-46. doi: 10.1016/j.jad.2025.02.047. Epub 2025 Feb 26. PMID 40021060
- [Derived] Kavakbasi E, Baune BT. Combination of Acute and Maintenance Esketamine Treatment With Adjunctive Long-Term Vagus Nerve Stimulation in Difficult-to-Treat Depression. Neuromodulation. 2024 Jun;27(4):766-773. doi: 10.1016/j.neurom.2023.12.004. Epub 2024 Feb 10. PMID 38340111
- [Derived] Kavakbasi E, Rosemann K, Yilmaz M, Vasileiadou A, Falcone V, Baune BT. Vagus Nerve Stimulation Combined With Alternating Synchronized and Nonsynchronized Intermittent Theta Burst Stimulation in Difficult-to-Treat Depression. J ECT. 2024 Mar 1;40(1):62-63. doi: 10.1097/YCT.0000000000000964. Epub 2023 Dec 28. No abstract available. PMID 38194603
- [Derived] Young AH, Juruena MF, De Zwaef R, Demyttenaere K. Vagus nerve stimulation as adjunctive therapy in patients with difficult-to-treat depression (RESTORE-LIFE): study protocol design and rationale of a real-world post-market study. BMC Psychiatry. 2020 Sep 29;20(1):471. doi: 10.1186/s12888-020-02869-6. PMID 32993573